CLINICAL TRIAL: NCT01130402
Title: A Real-time and Computerized Sonographic Scoring System for Predicting Malignant Cervical Lymphadenopathy
Brief Title: A Real-time and Computerized Sonographic Reporting System in Predicting Malignant Cervical Lymphadenopathy
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Research Ethics Review Committee, Far Eastern Memorial Hospital, Taipei, Taiwan
Other Study IDs: 098026-3
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2009-04

CONDITIONS: Lymphadenopathy
Keywords: age; lymphadenopathy; fine needle aspiration; sonography
MeSH Terms: conditions — Lymphadenopathy

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Neck masses: Patients with previously untreated neck masses

SUMMARY:
The investigaotors want to establish a real-time and computerized score reporting system based on the significant predictors of the measured sonographic parameters and demographic data.

DETAILED DESCRIPTION:
One hundred eight patients with neck lymphadenopathy, receiving ultrasonography and ultrasound-guided fine-needle aspiration (US-FNA), were used to construct a predictive model. This model was validated by another independent patient cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously untreated neck masses underwent neck US

Exclusion Criteria:

* The neck mass was not lymph node
* No US-FNA cytology result

Ages: 10 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with previously untreated neck masses were referred for sonographic evaluation and subsequent US-FNA after informed consent was obtained. Demographic data, including age and sex, side, site, and number of lymphadenopathy was collected as well.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2009-06; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The final diagnoses of lymph nodes were made by US-FNA cytological studies, pathologic results of the biopsy specimens, or at least 3 months of negative follow-up observations. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Li-Jen Liao, MD, Study Director — Department of Otolaryngology, Far Eastern Memorial Hospital, Taipei, Taiwan
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Liao LJ, Wang CT, Young YH, Cheng PW. Real-time and computerized sonographic scoring system for predicting malignant cervical lymphadenopathy. Head Neck. 2010 May;32(5):594-8. doi: 10.1002/hed.21225. PMID 19693943